CLINICAL TRIAL: NCT02797093
Title: Impact of ART Adherence on HIV Persistence and Inflammation
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 15-2309; 1R21AI124859-01 (NIH)
Record Dates: First submitted 2016-06-02; First posted 2016-06-13 (Estimated); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Human Immunodeficiency Virus
Keywords: anti-retroviral therapy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — The aim of the study is to quantify levels of CA-RNA, CA-DNA, and plasma residual viremia in suppressed, HIV infected individuals and correlate them with levels of TFV-DP in DBS as a measure of cumulate drug exposure (adherence). Second, the investigators will evaluate the changes in the HIV reservoir in relation to changes in ART adherence over time.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV suppressed individuals: HIV suppressed individuals on chronic ART, suboptimal adherence and exposure, measured through TFV-DP in DBS.

SUMMARY:
The purpose of this study is to evaluate the relationship between anti-retroviral therapy (ART) adherence with levels of human immunodeficiency virus (HIV) reservoir and residual viremia in suppressed, HIV-infected individuals on chronic ART.

DETAILED DESCRIPTION:
Understanding whether the size and dynamics of the HIV reservoir are associated with adherence, measured by an objective biomarker, could have significant clinical and therapeutic implications for ART and HIV cure.

1. First, this aim will quantify levels of CA-RNA, CA-DNA, and plasma residual viremia in suppressed, HIV infected individuals and correlate them with levels of TFV-DP in DBS as a measure of cumulate drug exposure (adherence).
2. Second, this study will evaluate the changes in the HIV reservoir in relation to changes in ART adherence over time.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-infected males and females,
2. Ages 18 years and older,
3. Taking any TFV-based regimen,
4. HIV suppression <20 copies/ml for at least 12 months;
5. Not co-infected with HCV;
6. Able and willing to give informed consent.

Exclusion Criteria:

1. Pregnancy.
2. Refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected individuals who are being treated with a tenofovir-based regimen.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2016-01; Primary Completion 2018-10-12 (Actual); Study Completion 2018-10-12 (Actual)

PRIMARY OUTCOMES:
Level of tenofovir diphosphate in dried blood spots associated with the size of the HIV reservoir measured by the amount of CA-RNA and CA-DNA in PBMCs. | 6 months
  Evaluation of variations in ART cumulative adherence are associated with the size of the HIV reservoir and with the degree of chronic inflammation and immune activation in HIV-infected, virologically suppressed individuals.

SECONDARY OUTCOMES:
Level of self-reported adherence (4-day, 30-day and 3-months using a visual analog scale) associated with the size of the HIV reservoir measured by CA-RNA and CA-DNA in PBMCs. | 6 months
  Evaluation of variations in ART self-reported adherence are associated with the size of the HIV reservoir and with the degree of chronic inflammation and immune activation in HIV-infected, virologically suppressed individuals.

CONTACTS AND LOCATIONS:
Overall Officials: Jose R Castillo-Mancilla, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No